CLINICAL TRIAL: NCT01087073
Title: Improving Diabetes Care and Outcomes on the South Side of Chicago
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16867B (TRACS ID: 40596); R18DK083946 (NIH); P30DK092949 (NIH); Alliance to Reduce Disparities (Other: Merck Company Foundation)
Record Dates: First submitted 2010-02-12; First posted 2010-03-15 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus
Keywords: Healthcare Disparities; Health Care Quality Improvement; Shared Decision-Making; Patient Education; Patient Activation; Community Outreach; Provider Training
MeSH Terms: conditions — Diabetes Mellitus; Patient Participation | interventions — Patient Education as Topic; Quality Improvement; Community-Institutional Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Patient Activation (Experimental): Patient knowledge in diabetes self-management behaviors and clinical measures (HbA1c, LDL, HDL, BMI, BP) are tracked at baseline, 10-weeks (post-program), 3 months (post-program) and 6 months (post-program).
  Interventions: Behavioral: Patient Activation
- Provider Training Evaluation (Experimental): Pre-post surveys are conducted at each training session to assess overall satisfaction with the curriculum, knowledge of SDM, and understanding of techniques to promote its use in the healthcare setting.
  Interventions: Behavioral: Provider Training
- Quality Improvement Evaluation (Experimental): We measure quality improvement efforts through biannual staff experience surveys and one-on-one provider and clinic staff interviews.
  Interventions: Behavioral: Quality Improvement
- Community Outreach Evaluation (Experimental): Pre-post surveys will be disseminated at nutrition tours (Save-A-Lot, Walgreens, 61st Street Farmers Market) to assess change in knowledge of healthy eating behaviors and proper nutrition. Surveys will also assess participant satisfaction of the tours.
  Interviews will also be performed with community stakeholders to assess the costs/benefits of the collaboration and overall feedback on involvement.
  Interventions: Behavioral: Community Outreach
- Global Evaluation of the Intervention (No Intervention): A chart review will be performed in order to evaluate our intervention to improve diabetes processes of care and clinical outcomes among our target population. Chart abstractions will be performed on medical records obtained from our six intervention clinics. In addition, chart abstractions from two University of Illinois at Chicago clinics and three FQHCs located on the West Side of Chicago will serve as control data.100 charts will be randomly selected from each clinic per year of the intervention. The chart review will contain charts from adult diabetes patients over a seven year period that matches the duration of the Improving Diabetes project.

INTERVENTIONS:
Behavioral: Patient Activation — Culturally tailored patient activation training classes providing education and communication strategies to empower patients to be proactive in their diabetes self-management behavior. Participants attend a 10 week interactive class. Diabetes support groups after the completion of these classes help patient maintain self-management and adherence to healthy behaviors.
  Other Names: Patient Education
  Arms: Patient Activation
Behavioral: Provider Training — Provider patient-centered communication training focuses on cultural competency and communication skills training to aid in shared decision-making and tailoring treatment recommendations to the patient's cultural preferences and readiness. Providers attend 4 1-hour monthly modules and one booster workshop 3 months post-class.
  Arms: Provider Training Evaluation
Behavioral: Quality Improvement — Participating clinics participate in quality improvement (QI) programs which aim to redesign clinic operations to improve care for diabetes patients. QI initiatives have included instituting group visits, patient medication cards, peer support groups, flow sheets, nurse case management, and patient registries. New initiatives include improving access and tracking of specialists visits, employing community health workers/patient navigators, coordinating care, and implementing other team-based care initiatives. Provider and clinical staff members from all six project clinics attend collaborative quarterly QI sessions with project staff to discuss improvements in QI efforts, share QI methods among clinic teams, and provide brief training sessions.
  Arms: Quality Improvement Evaluation
Behavioral: Community Outreach — The project collaborates with many community based organizations and resources to reach out to communities at high risk for diabetes on the South Side of Chicago and facilitate diabetes education, particularly in the area of nutrition and physical activity. We provide monthly health education events, nutrition tours, and frequently participate in community-based health fairs and health promotion events. We also work to promote nutrition through the Food Rx program, which utilizes a prescription to link patients at our clinics with nutrition resources on the South Side of Chicago through a coupon that gives discounts towards healthy purchases at participating stores, and have initiated a 10-week fitness program to promote physical activity among minority patients with diabetes.
  Other Names: Community Partnerships
  Arms: Community Outreach Evaluation

SUMMARY:
The Improving Diabetes Care and Outcomes project aims to reduce diabetes disparities and engages patients, providers, clinics, and community collaborators to improve the health care and outcomes of African-Americans on the South Side of Chicago. Initiated in 2009, this project is a collaborative, community-based intervention that employs a multifaceted, integrated approach to address many of the root causes of health disparities. The short-term goal of this project is to improve clinic processes such as appointment scheduling and patient counseling through quality improvement efforts, as well as clinical outcomes including HbA1c, cholesterol and blood pressure in patients with diabetes through patient education. Long-term goals are to strengthen the network of community health centers, community-based organizations and academic medical centers, while increasing awareness of local diabetes disparities and empowering communities to combat this problem.

DETAILED DESCRIPTION:
This multifactorial intervention contains four overlapping core components reflecting key elements of the Chronic Care Model.This model identifies patients, practice teams, the community, and health systems as four necessary elements in the successful management of chronic diseases such as diabetes. Six health centers (two academic center clinics affiliated with the University of Chicago and four FQHCs) are part of the intervention. Researchers at the University of Chicago received grant funding from the Merck Company Foundation's Alliance to Reduce Disparities in Diabetes and the National Institutes of Health to implement and evaluate the intervention.

The research and implementation team includes faculty and staff members with expertise in quality improvement, behavioral change, community outreach, patient education, and research methods.

The intervention has four main components:

1. Patient Activation: We hold culturally tailored, 10-week patient education classes that combine culturally tailored patient education with training in shared decision-making skills to empower patients to be proactive in their diabetes self-management.
2. Provider Training: We provide educational workshops for provider, clinical, and non-clinical staff at our six intervention clinics on patient-centered communication, cultural competency, behavior change counseling, and shared decision making.
3. Quality Improvement: Our team facilitates quality improvement (QI) programs redesigning clinic operations to improve care for diabetes patients. QI initiatives have included instituting group visits, patient medication cards, peer support groups, flow sheets, nurse case management, and patient registries. New initiatives include improving access and tracking of specialists visits through EMR, employing community health workers/patient navigators, coordinating care, and implementing other team-based care initiatives. We also perform a cost/benefits analysis of intervention implementation from the business case perspective of the outpatient clinics and determine the major barriers and solutions to successfully implement and sustain the project at each location.
4. Community Outreach: We collaborate with existing community resources to create sustainable collaborations that support diabetes patients outside of the health care system and promote nutrition and a healthy lifestyle. We collaborate with grocery stores, food pantries, the Chicago Park District, farmers markets, media outlets, grocery stores and other community-based organizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diabetes diagnosis (ICD-9 codes 250.X) and be age 18 years or older
* Patients must attend one of the participating health centers

Exclusion Criteria:

* Gestational diabetes patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6209 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline data will be collected at the end of 1st year; follow-up data will be collected from years 2-7.
  Chart audit will be conducted on 100 randomly selected diabetes patients meeting the age inclusion criteria (age 18 years and older). Will also be collected from patients in the patient activation component.
Blood pressure | Baseline data will be collected at the end of 1st year; follow-up data will be collected from years 2-7.
  Chart audit will be conducted on 100 randomly selected diabetes patients meeting the age inclusion criteria (age 18 years and older). Will also be collected from patients in the patient activation component.
Lipids (HDL, LDL, total cholesterol, triglycerides) | Baseline data will be collected at the end of 1st year; follow-up data will be collected from years 2-7.
  Chart audit will be conducted on 100 randomly selected diabetes patients meeting the age inclusion criteria (age 18 years and older). Will also be collected from patients in the patient activation component.

SECONDARY OUTCOMES:
Processes of care | Baseline data will be collected at the end of 1st year; follow-up data will be collected from years 2-7.
  Chart audit will be conducted on 100 randomly selected diabetes patients meeting the age inclusion criteria (age 18 years and older).
  Annual Processes of Care:
  At least 1 HbA1c, Lipid assessment, Microalbumin assessment, ACE inhibitor or ARB prescribed, Aspirin prescribed, Dental referral, Eye exam or referral, Foot exam or referral, Influenza vaccination, Home glucose monitoring, Dietary counseling or referral, Exercise counseling, Diabetes education

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Chin, MD, MPH, Principal Investigator — University of Chicago; Monica Peek, MD, MPH, Principal Investigator — University of Chicago
Locations (6):
- United States (6):
  - ACCESS Grand Boulevard Family Health Center, Chicago, Illinois
  - Friend Family Health Center, Chicago, Illinois
  - Chicago Family Health Center, Chicago, Illinois
  - Kovler Diabetes Center, Chicago, Illinois
  - University of Chicago, Primary Care Group, Chicago, Illinois
  - ACCESS Booker Family Health Center, Chicago, Illinois

REFERENCES:
- [Background] Peek ME, Ferguson M, Bergeron N, Maltby D, Chin MH. Integrated community-healthcare diabetes interventions to reduce disparities. Curr Diab Rep. 2014 Mar;14(3):467. doi: 10.1007/s11892-013-0467-8. PMID 24464339
- [Background] Wilkes AE, Bordenave K, Vinci L, Peek ME. Addressing diabetes racial and ethnic disparities: lessons learned from quality improvement collaboratives. Diabetes Manag (Lond). 2011 Nov;1(6):653-660. doi: 10.2217/dmt.11.48. PMID 22563350
- [Background] Nundy S, Lu CY, Hogan P, Mishra A, Peek ME. Using Patient-Generated Health Data From Mobile Technologies for Diabetes Self-Management Support: Provider Perspectives From an Academic Medical Center. J Diabetes Sci Technol. 2014 Jan;8(1):74-82. doi: 10.1177/1932296813511727. Epub 2014 Jan 1. PMID 24876541
- [Background] Nundy S, Dick JJ, Chou CH, Nocon RS, Chin MH, Peek ME. Mobile phone diabetes project led to improved glycemic control and net savings for Chicago plan participants. Health Aff (Millwood). 2014 Feb;33(2):265-72. doi: 10.1377/hlthaff.2013.0589. PMID 24493770
- [Background] Nundy S, Dick JJ, Solomon MC, Peek ME. Developing a behavioral model for mobile phone-based diabetes interventions. Patient Educ Couns. 2013 Jan;90(1):125-32. doi: 10.1016/j.pec.2012.09.008. Epub 2012 Oct 10. PMID 23063349
- [Background] Nundy S, Dick JJ, Goddu AP, Hogan P, Lu CY, Solomon MC, Bussie A, Chin MH, Peek ME. Using mobile health to support the chronic care model: developing an institutional initiative. Int J Telemed Appl. 2012;2012:871925. doi: 10.1155/2012/871925. Epub 2012 Dec 5. PMID 23304135
- [Background] Peek ME, Gorawara-Bhat R, Quinn MT, Odoms-Young A, Wilson SC, Chin MH. Patient trust in physicians and shared decision-making among African-Americans with diabetes. Health Commun. 2013;28(6):616-23. doi: 10.1080/10410236.2012.710873. Epub 2012 Oct 10. PMID 23050731
- [Background] Peek ME, Tang H, Cargill A, Chin MH. Are there racial differences in patients' shared decision-making preferences and behaviors among patients with diabetes? Med Decis Making. 2011 May-Jun;31(3):422-31. doi: 10.1177/0272989X10384739. Epub 2010 Dec 2. PMID 21127318
- [Background] Peek ME, Wagner J, Tang H, Baker DC, Chin MH. Self-reported racial discrimination in health care and diabetes outcomes. Med Care. 2011 Jul;49(7):618-25. doi: 10.1097/MLR.0b013e318215d925. PMID 21478770
- [Background] Peek ME, Odoms-Young A, Quinn MT, Gorawara-Bhat R, Wilson SC, Chin MH. Race and shared decision-making: perspectives of African-Americans with diabetes. Soc Sci Med. 2010 Jul;71(1):1-9. doi: 10.1016/j.socscimed.2010.03.014. Epub 2010 Mar 24. PMID 20409625
- [Background] Peek ME, Odoms-Young A, Quinn MT, Gorawara-Bhat R, Wilson SC, Chin MH. Racism in healthcare: Its relationship to shared decision-making and health disparities: a response to Bradby. Soc Sci Med. 2010 Jul;71(1):13-7. doi: 10.1016/j.socscimed.2010.03.018. Epub 2010 Mar 24. No abstract available. PMID 20403654
- [Background] Chin MH, Walters AE, Cook SC, Huang ES. Interventions to reduce racial and ethnic disparities in health care. Med Care Res Rev. 2007 Oct;64(5 Suppl):7S-28S. doi: 10.1177/1077558707305413. PMID 17881624
- [Background] Peek ME, Cargill A, Huang ES. Diabetes health disparities: a systematic review of health care interventions. Med Care Res Rev. 2007 Oct;64(5 Suppl):101S-56S. doi: 10.1177/1077558707305409. PMID 17881626
- [Background] Chin MH. Quality improvement implementation and disparities: the case of the health disparities collaboratives. Med Care. 2010 Aug;48(8):668-75. doi: 10.1097/MLR.0b013e3181e3585c. PMID 20613665
- [Result] Raffel KE, Goddu AP, Peek ME. "I Kept Coming for the Love": Enhancing the Retention of Urban African Americans in Diabetes Education. Diabetes Educ. 2014 May;40(3):351-360. doi: 10.1177/0145721714522861. Epub 2014 Feb 13. PMID 24525568
- [Result] Peek ME, Wilkes AE, Roberson TS, Goddu AP, Nocon RS, Tang H, Quinn MT, Bordenave KK, Huang ES, Chin MH. Early lessons from an initiative on Chicago's South Side to reduce disparities in diabetes care and outcomes. Health Aff (Millwood). 2012 Jan;31(1):177-86. doi: 10.1377/hlthaff.2011.1058. PMID 22232108
- [Result] Peek ME, Harmon SA, Scott SJ, Eder M, Roberson TS, Tang H, Chin MH. Culturally tailoring patient education and communication skills training to empower African-Americans with diabetes. Transl Behav Med. 2012 Sep;2(3):296-308. doi: 10.1007/s13142-012-0125-8. PMID 24073128
- [Result] Chin MH, Goddu AP, Ferguson MJ, Peek ME. Expanding and sustaining integrated health care-community efforts to reduce diabetes disparities. Health Promot Pract. 2014 Nov;15(2 Suppl):29S-39S. doi: 10.1177/1524839914532649. PMID 25359247
- [Result] Peek ME, Ferguson MJ, Roberson TP, Chin MH. Putting theory into practice: a case study of diabetes-related behavioral change interventions on Chicago's South Side. Health Promot Pract. 2014 Nov;15(2 Suppl):40S-50S. doi: 10.1177/1524839914532292. PMID 25359248
- See also: Improving Diabetes Care and Outcomes Project Website — http://southsidediabetes.com/